CLINICAL TRIAL: NCT05304052
Title: Mindful Awareness Practices vs. Wait List Control Randomized Controlled Trial for College Students: Effects on Psychosocial Outcomes and Neural and Immune Processes
Brief Title: Mindfulness Meditation Neuroimaging Study for Undergraduates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Julienne Bower, PhD, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-002038
Record Dates: First submitted 2022-02-09; First posted 2022-03-31 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Inflammation; Psychosocial Functioning; Depression, Anxiety
Keywords: adolescents; mindfulness meditation; brain imaging; inflammation
MeSH Terms: conditions — Inflammation; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: After completing the pre-intervention assessment (consisting of completing an online survey, a blood draw and brain scan while performing tasks in a fMRI machine), students will be randomized to one of the two study conditions. Study subjects will be informed of their assigned condition and those assigned to the mindfulness meditation class will be provided with specific details for the class, while those assigned to the wait list control group won't be expected to do anything during the six week class schedule, other than not to take any meditation classes.
Who Masked: Outcomes Assessor
Masking Description: Study coordinators who will be consenting and responsible for the pre-treatment and post-treatment assessments will be masked so that they will not have any bias as to which students participated in the mindfulness meditation intervention and which were in the wait list control group. A research associate who will not be participating in the assessments will be the one to call subjects and inform them of their assigned study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness meditation intervention (Experimental): Half of the subjects will be randomly assigned to participate in the mindfulness meditation intervention. This class will meet once a week, for two hours, over the course of six weeks.
  Interventions: Behavioral: Mindfulness Meditation classes
- Wait list control (No Intervention): Half of the subjects will be randomly assigned to be in the wait-list control group. These subjects will not be asked to do anything during the six weeks while the mindfulness meditation group takes place, other than to not enroll in a meditation class.

INTERVENTIONS:
Behavioral: Mindfulness Meditation classes — The mindful awareness practices (MAPS) intervention is based on an institutional program developed by the Mindful Awareness Research Center (MARC) at UCLA, but takes a more practical and accessible approach that focuses specifically on the practice of mindfulness and its application in everyday life (as compared to the focus on stress and stress reduction in mindfulness-based stress reduction). Key components of the intervention include development of bodily awareness, managing pain, working with difficult thoughts and feelings, cultivating positive emotions and loving kindness, and relational mindfulness practices. Each session provides structured training and exercises in mindfulness, including formal meditation practices and strategies for the daily informal use of mindfulness, as well as opportunity for group discussion and sharing. Participants will be instructed to practice mindfulness techniques on a daily basis, beginning with five minutes and increasing to 20 minutes.
  Arms: Mindfulness meditation intervention

SUMMARY:
This study is designed to test the effectiveness of mindfulness meditation intervention classes on psychosocial health outcomes. Additionally, the investigators would like to examine changes in the brain that might occur following the mindfulness meditation intervention. The investigators are particularly interested in changes in brain activity that are correlated with changes in inflammation-related markers in the blood. The nervous system and immune system are closely connected, and both are influenced by mindfulness. However, it is unclear whether changes in neural activity are linked with changes in inflammation. A compelling feature of mindfulness interventions is their potential for reducing inflammatory activity; however, this has not been examined in college students. In addition to measuring psychosocial outcomes, the investigators will employ sophisticated, vertically-integrated measures of inflammatory biology that allow the study team to probe intervention effects on circulating markers of inflammation.

Thus, the investigators intend to recruit 60 undergraduate students and will randomize them into either a 6-week standardized mindfulness intervention or to a wait-list control group. Participants will complete brain scans, provide blood samples for immune analysis, and complete questionnaires at pre- and post-intervention assessments

DETAILED DESCRIPTION:
Psychosocial symptoms, such as depression and anxiety, are often elevated in adolescents, particularly as they transition to college. Mental health stress can also lead to negative effects in underlying biological markers of health, such as inflammation. Inflammation is linked to alterations in emotion, cognitive function, and behavior, and is increasingly recognized as a key contributor to mental and physical health.

Mindfulness-based interventions (MBIs) offer a promising alternative for addressing psychosocial symptoms among college students. Mindfulness involves bringing attention to one's present moment experiences, including thoughts, feelings, and physical sensations, with openness, curiosity, and absence of judgment. Interventions have been developed to cultivate mindfulness through formal meditation and informal practice, and RCTs (randomized controlled trials) have documented benefits of mindfulness-based interventions on psychological and biological health outcomes.

The UCLA Mindful Awareness Research Center (MARC) has developed and validated a group-based mindfulness intervention, Mindful Awareness Practices (MAPs), that has demonstrated beneficial effects on mental health in adults and may offer a promising, scalable approach for improving associated psychological and biological outcomes in college students. More rigorous evaluation among college students, relative to a wait list control condition, is required for validation and before broad implementation of this promising approach can occur.

Overview: The proposed randomized controlled trial (RCT) will investigate the effect of a standardized mindfulness intervention on psychological, neural, and inflammatory processes in college students compared to a wait list control group. Furthermore, the investigators will examine the association between changes in psychological, neural, and immune outcomes.

Participants: Study participants will be undergraduate students at the University of California, Los Angeles (UCLA). They will be recruited in cohorts of 30 and randomized 1:1 to one of the two study arms (15 students in MAPs class/15 wait list control). Participants will complete online questionnaires, a functional magnetic resonance imaging (fMRI) scan and will provide blood samples before and after the six-week intervention period.

Screening: Potential subjects will be screened for eligibility over the phone. The 4-item Patient Health Questionnaire (PHQ4) will be administered to assess mood (depression and anxiety). If a potential subject scores a "3" on either subscale, the study coordinator will administer the 8-item Patient Health Questionnaire (PHQ8)(for depression) or the GAD-7 (for anxiety) to determine the severity. If the potential participant scores "15" or more on either scale, they will be referred to the UCLA Counseling and Psychological Services (CAPS).

Enrollment and Baseline Assessment (T1): All students who are determined to be eligible will be scheduled for an in-person, baseline assessment (T1) at the UCLA Health Psychology Laboratory (HPL). The Institutional Review Board (IRB) approved consent form will be reviewed and signed. A pre-intervention online survey will also be completed during this initial in-person visit. The survey will consist of the following scales: Background demographic characteristics, health behaviors, Pittsburgh Sleep Quality Index (PSQI), Center for Epidemiological Studies-Depression (CES-D), Snaith-Hamilton Pleasure scale (SHAPS), Generalized Anxiety Disorder-7 (GAD-7), Perceived Stress Scale (PSS), UCLA Loneliness Scale, Positive and Negative affect (PANAS-X), Mental Health Continuum-short form, Mindfulness scale (FFMQ), Self-compassion scale, Rumination and reflection questionnaire, Ways of Savoring checklist (WOSC), Compassion scale and the Tennessee Self-concept short form scale (TSCS) .

Participants will provide blood samples for immune evaluation. Due to changes in research procedures due to COVID-19, the investigators would like to change the usual method for blood collection. Prior to COVID-19, blood was drawn by venipuncture by a licensed phlebotomist. However, in order to mitigate risk and abide to social distancing guidelines. the investigators now plan to collect blood by utilizing the Tasso OnDemand device, which allows self-collection of a single capillary blood sample and does not require venipuncture. The Tasso device sticks to the skin with a light adhesive. When the button is pressed, a vacuum forms and a lancet pricks the surface of the skin. The vacuum draws blood out of the capillaries and into a sample pod attached to the bottom of the device. The participant would watch a demonstration video during their baseline assessment visit, and then use the device to collect a blood sample. Approximately 1/8th of a teaspoon of blood will be drawn at each in-person assessment.

Subjects will also complete a 75 minute scan while lying in a fMRI machine. During the neuroimaging session, participants will undergo a series of probe tasks that are known to activate the neural regions of interest. In particular, the investigators will evaluate activity in the amygdala and related "neural alarm" regions in response to threat-related tasks, which the investigators hypothesize will decrease following mindfulness training. In addition, the investigators will examine activity in reward-related regions following compassion and self-affirmation tasks, which the investigators hypothesize will increase following mindfulness.

Baseline visits will be conducted in the 2-week period before intervention onset.

Randomization: After completing the baseline assessment, participants will be randomized to one of the two study conditions. The coordinator will inform the participants of their assigned condition and will provide information to those who will be taking the MAPs classes (the wait list control group won't be expected to do anything during the six week class schedule, other than not to take any meditation classes).

Intervention: Mindful Awareness Practices (MAPs): Participants assigned to this condition will be asked to attend two-hour group sessions once a week for six weeks. The MAPs intervention is based on an institutional program developed by the Mindful Awareness Research Center (MARC) at UCLA. The MAPs program is similar to other mindfulness-based interventions in its general focus on cultivating mindfulness, but takes a more practical and accessible approach that focuses specifically on the practice of mindfulness and its application in everyday life (as compared to the focus on stress and stress reduction in mindfulness-based stress reduction). Key components of the intervention include development of bodily awareness, managing pain, working with difficult thoughts and feelings, cultivating positive emotions and loving kindness, and relational mindfulness practices. Each session provides structured training and exercises in mindfulness, including formal meditation practices and strategies for the daily informal use of mindfulness, as well as opportunity for group discussion and sharing. Home practice is a key component of MAPs. Participants will be instructed to practice mindfulness techniques on a daily basis, beginning with five minutes and increasing to 20 minutes. Subjects will be asked to complete daily homework logs throughout the 6-weeks.

The MAPs curriculum will be implemented by trained instructors who will receive specialized training in delivery of the study-specific protocol and will be overseen by Dr. Marvin Belzer, Associate Director of the MARC and master instructor for this trial. MAPs classes will be held in private rooms in the residential part of the UCLA campus, close to student living quarters. MAPs classes will be conducted in the evenings and scheduled to occur mid-way through the quarter to minimize conflict with classes and exam periods.

Immediate Post-Intervention Assessment (T2): This in-person visit will be scheduled to occur within 2 weeks after the conclusion of the study interventions at the UCLA Health Psychology Lab and will include completion of a post-intervention online questionnaire (all scales from the baseline will be administered again except for the demographic characteristics), collection of blood samples using the TASSO OnDemand device (approximately 1/8 teaspoon), and another 75 minute fMRI neuroimaging session.

After the post-intervention assessments have been completed, students who were assigned to the wait-list control group will be offered the opportunity to take the MAPs class.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students at UCLA
* Must live on the UCLA campus
* Must be right-handed (for the fMRI scan)

Exclusion Criteria:

* Current diagnosis of mood or anxiety disorder as determined by the PHQ-8 or by the GAD-7 if score "15" or more on either measure
* Presence of medical conditions or use of medications that may influence inflammation (e.g., autoimmune disorder)
* Regular tobacco use
* Actively practicing mindfulness meditation
* Left-handed (for the fMRI scan)
* BMI > 30 (for the fMRI scan)
* Pregnant (for the fMRI scan)
* Color blind (for the fMRI scan)
* Non-removable metal in body (for the fMRI scan)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-03-27 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Psychological well-being | Baseline and at 8 weeks
  Change in psychological well-being
  Well-being will be measured via the 14-item Mental Health Continuum-Short Form (MHC-SF). The MHC-SF is comprised of three empirically derived subscales: the 3-item Emotional Well-Being Subscale, the 6-item Psychological Well-Being Subscale, and the 5-item Social Well-Being Subscale. Higher scores on each subscale, and the total score overall (range: 0-56), indicate greater well-being.
Depression | Baseline and at 8 weeks
  Change in depressive symptoms
  Depressive symptoms will be measured via the 20-item Center for Epidemiological Studies Depression Scale (CES-D). The CES-D is a measure of symptom severity, with higher scores (range: 0-60) indicating greater depressive symptoms
Anxiety | Baseline and at 8 weeks
  Change in anxiety
  Symptoms of anxiety will be measured via the 7-item Generalized Anxiety Disorder- 7 (GAD-7). Higher scores on the GAD-7 (range: 0-21) indicate greater severity of symptoms.
Perceived stress | Baseline and at 8 weeks
  Change in perceived stress Perceived stress will be measured via the 10-item Perceived Stress Scale (range: 0-40). Higher scores indicate greater perceived stress levels.

SECONDARY OUTCOMES:
Inflammation | Baseline and at 8 weeks
  The primary immune outcome of interest is inflammatory gene expression, measured through a set of 19 pre-specified pro-inflammatory gene transcripts that have previously been shown to be upregulated in the context of chronic stress and downregulated by the mindfulness meditation intervention. The inflammatory composite includes the following genes: IL1A, IL1B, IL6, IL8, TNF, PTGS1, PTGS2, FOS, FOSB, FOSL1, FOSL2, JUN, JUNB, JUND, NFKB1, NFKB2, REL, RELA, and RELB)
Mindfulness | Baseline and at 8 weeks
  Change in Mindfulness
  Mindfulness will be measured via the 39-item Five Facet Mindfulness Questionnaire (FFMQ). The FFMQ has both direct and reverse scoring items and is comprised of 5 subscales: observing, describing, acting with awareness, non-judgment and non-reactivity, along with an overall mindfulness score. The total FFMQ can be divided by 39 to get an average item score. Scores represent a spectrum of mindfulness.
Positive and negative affect | Baseline and at 8 weeks
  Change in positive and negative affect
  Reports of positive and negative affect will be assessed via the 10-item positive affect subscale and 10-item negative affect subscales of the Positive and Negative Affect Schedule (PANAS-X). Two additional adjectives were also included, happy and calm. Greater scores indicate higher feelings of positive (range: 10-50) and negative affect (range: 10-50).
Anhedonia | Baseline and at 8 weeks
  Change in anhedonia
  Anhedonia will be measured via the 14-item Snaith-Hamilton Pleasure Scale which covers domains of social interaction, food and drink, sensory experiences and interests/pastimes. Scores range from 0-14 with higher scores indicating the inability to experience pleasure.
Loneliness | Baseline and at 8 weeks
  Change in loneliness
  Loneliness will be measured via the 3-item UCLA Loneliness Scale (range: 3-9). Higher scores indicate greater loneliness
Rumination | Baseline and at 8 weeks
  Change in Rumination
  Rumination will be measured via the 6-item rumination subscale from the Rumination and Reflection questionnaire. Some items require reverse scoring. Rumination reflects a tendency to focus on negative self-perceptions.
Compassion for others | Baseline and at 8 weeks
  Change in compassion for others Compassion for others will be measured via the 16-item Compassion scale. This measure contains four subscales: greater kindness, common humanity, mindfulness and lessened indifference. Some items are reverse scored. Each scale is scored by taking the mean.
Sleep disruption (sleep latency, sleep duration, sleep efficiency, sleep disturbance and daytime dysfunction) | Baseline and at 8 weeks
  Changes in sleep disruption will be examined by looking at changes in sleep latency, sleep duration, sleep efficiency, sleep disturbance and daytime dysfunction.
  Sleep disruption will be measured via the Pittsburgh Sleep Quality Index. 19 self-rated items are combined to form seven "component" scores, (sleep latency, sleep duration, sleep efficiency, sleep disturbance, daytime dysfunction, with subjective sleep quality rated by participant, and use of sleep medications included in scale) each of which ranges from 0-3 points ("0 indicates no difficulty, while "3" indicates severe difficulty). The seven component scores are combined into one "global" score, ranging from 0-21 points. Higher scores indicate greater sleep disruption.
Savoring strategies | Baseline and at 8 weeks
  Change in savoring strategies
  The degree to which people engage in savoring strategies will be measured via the 60-item Ways of Savoring Checklist (WOSC) scale. This measure contains three subscales of interest when it comes to mindfulness: absorption, temporal awareness, and kill-joy thinking items. Some items are reverse scored. Each scale is scored by taking the mean.
Self-concept | Baseline and at 8 weeks
  Change in self-concept Self-concept will be measured via the 20-item Tennessee Self-concept short form scale (TSCS-SF). This short form version measures total self-concept with higher scores indicating greater strength in one's self-view.
Self-compassion | Baseline and at 8 weeks
  Change in self-compassion
  Self-compassion will be measured via the 26-item Self-compassion scale. This scale contains 6 subscales: self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification. Subscale scores are computed by calculating the mean of subscale item responses or a total self-compassion score can be computed after reverse scoring the negative subscale items and then computing a mean. There are no clinical scores which indicate that an individual is high or low in self-compassion. Rather, scores are often used in a comparative manner to examine outcomes for people who score either higher or lower in self-compassion.

CONTACTS AND LOCATIONS:
Overall Officials: Julienne E Bower, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share any individual participant data (IPD) with any other researchers. Data will be reported in group form to prevent personal identification of participants. When the research has been completed, the data will be stored in a secured area of a private, locked research office. Any personal identifiers and/or codes linking the data to personal identifiers will be kept on a separate computer with password protection for reference and for future research. All personal identifiers will be kept confidential. Only identified members of the research team and the P.I. will have access to the data, identifiers and/or codes. Data with subject identifiers will not be released to any agency or persons.